CLINICAL TRIAL: NCT04472650
Title: A Phase 1, Open-label, Single-dose, Randomized Crossover Study to Evaluate the Relative Bioavailability of Two Different Capsule Formulations of Sitravatinib in Healthy Subjects
Brief Title: Relative Bioavailability of Two Different Capsule Formulations of Sitravatinib in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: BeiGene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: BGB-Sitravatinib-101
Record Dates: First submitted 2020-07-14; First posted 2020-07-15 (Actual); Results first posted 2021-12-27 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Tumor
MeSH Terms: conditions — Neoplasms | interventions — sitravatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Dosing Sequence 1: Sitravatinib Free Base then Malate Salt (Experimental): Sitravatinib free base capsule 120 mg on Day 1 in Period 1 then sitravatinib malate salt capsule 100 mg on Day 1 in Period 2, with a minimum washout period between dose administrations of 14 days
  Interventions: Drug: Sitravatinib
- Dosing Sequence 2: Sitravatinib Malate Salt then Free Base (Experimental): Sitravatinib malate salt capsule 100 mg on Day 1 in Period 1 then sitravatinib free base capsule 120 mg on Day 1 in Period 2, with a minimum washout period between dose administrations of 14 days
  Interventions: Drug: Sitravatinib

INTERVENTIONS:
Drug: Sitravatinib — Administered orally as a free base capsule
Drug: Sitravatinib — Administered orally as a malate salt capsule

SUMMARY:
The primary objective of the study was to investigate the relative bioavailability and pharmacokinetics (PK) of sitravatinib free base and malate salt capsule formulations following oral administration in healthy adults.

ELIGIBILITY:
Key Inclusion Criteria:

1. Body mass index between 18.0 and 32.0 kg/m2, inclusive.
2. In good health, determined by no clinically significant findings from medical history, physical examination, 12-lead ECG, vital sign measurements, and clinical laboratory evaluations at Screening and/or Check-in as assessed by the Investigator (or designee).
3. Able to swallow multiple capsules.

Key Exclusion Criteria:

1. History of stomach or intestinal surgery or resection
2. Have previously completed or withdrawn from this study or any other study investigating sitravatinib and have previously received the investigational product.
3. Participants who, in the opinion of the Investigator (or designee), should not participate in this study.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2020-07-23 (Actual); Primary Completion 2020-11-09 (Actual); Study Completion 2020-11-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Principal Investigator — BeiGene
Locations (1):
- Linear Clinical Research, Nedlands, Western Australia, Australia

IPD SHARING:
Plan to Share IPD: Yes

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were randomized in a 1:1 ratio in two dosing sequences in a 2-period crossover design at a single site in Australia. Periods 1 and 2 were separated by a minimum of 14 days between dose administrations. Total duration of study participation was up to approximately 8 weeks.
Groups:
- Dosing Sequence 1: Sitravatinib Free Base Capsule Then Malate Salt Capsule: Sitravatinib free base capsule 120 mg on Day 1 of Period 1 then sitravatinib malate salt capsule 100 mg on Day 1 of Period 2, with a minimum washout period between dose administrations of 14 days
- Dosing Sequence 2: Sitravatinib Malate Salt Capsule Then Free Base Capsule: Sitravatinib malate salt capsule 100 mg on Day 1 of Period 1 then sitravatinib free base capsule 120 mg on Day 1 of Period 2, with a minimum washout period between dose administrations of 14 days
Period: Period 1 (Up to 15 Days)
Arm/Group | Dosing Sequence 1: Sitravatinib Free Base Capsule Then Malate Salt Capsule | Dosing Sequence 2: Sitravatinib Malate Salt Capsule Then Free Base Capsule
Started | 13 | 13
Completed | 13 | 13
Not Completed | 0 | 0
Period: Washout Period (Minimum 14 Days)
Arm/Group | Dosing Sequence 1: Sitravatinib Free Base Capsule Then Malate Salt Capsule | Dosing Sequence 2: Sitravatinib Malate Salt Capsule Then Free Base Capsule
Started | 13 | 13
Completed | 12 | 13
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0
Period: Period 2 (Up to 15 Days)
Arm/Group | Dosing Sequence 1: Sitravatinib Free Base Capsule Then Malate Salt Capsule | Dosing Sequence 2: Sitravatinib Malate Salt Capsule Then Free Base Capsule
Started | 12 | 13
Completed | 12 | 13
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set included participants who received at least 1 dose of sitravatinib
Groups:
- Total: Total of all reporting groups
Arm/Group | Dosing Sequence 1: Sitravatinib Free Base Capsule Then Malate Salt Capsule | Dosing Sequence 2: Sitravatinib Malate Salt Capsule Then Free Base Capsule | Total
Number analyzed (Participants) | 13 | 13 | 26
Age, Continuous [Mean (Standard Deviation); unit: Years] | 27.1 (4.23) | 28.2 (10.19) | 27.7 (7.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 13 | 13 | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 13 | 13 | 26
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 8 | 9 | 17
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 2 | 0 | 2
  White | 3 | 3 | 6
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration-time Curve (AUC) From Time Zero to Infinity (AUC0-∞) of Sitravatinib
Time Frame: Predose and 0.5, 1, 2, 4, 6, 8, 12, 24, 48, 72 and 168 hours postdose in each study period
Population: Pharmacokinetic (PK) parameters analysis set included all participants who received at least 1 dose of sitravatinib and had at least 1 PK parameter of sitravatinib
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Groups:
- Sitravatinib Malate Salt Capsule: Sitravatinib malate salt capsule 100 mg (test) on Day 1 of Periods 1 and 2, with a minimum washout period between dose administrations of 14 days
- Sitravatinib Free Base Capsule: Sitravatinib free base capsule 120 mg (reference) on Day 1 of Periods 1 and 2, with a minimum washout period between dose administrations of 14 days
Arm/Group | Sitravatinib Malate Salt Capsule | Sitravatinib Free Base Capsule
Number analyzed (Participants) | 25 | 26
h*ng/mL | 2524.7 (28.8) | 2892.6 (34.5)
Statistical Analysis 1: Comparison: Sitravatinib Malate Salt Capsule vs Sitravatinib Free Base Capsule; Sitravatinib Malate Salt Capsule (Test) vs. Sitravatinib Free Base Capsule (Reference). Analysis based on Relative Bioavailability Analysis Set, defined as the subset of participants in the PK Parameters Analysis Set who had at least 1 primary PK parameter (AUC0-t, AUC0-inf and Cmax of sitravatinib) in both periods; Test type: Other; Ratio of Geometric Least Squares Means = 87.63, 90% CI 2-sided [78.273 to 98.111]

2. Primary Outcome: Area Under the Concentration-time Curve From Time Zero to Time of the Last Quantifiable Concentration (AUC0-t) of Sitravatinib
Time Frame: Predose and 0.5, 1, 2, 4, 6, 8, 12, 24, 48, 72 and 168 hours postdose in each study period
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Sitravatinib Malate Salt Capsule | Sitravatinib Free Base Capsule
Number analyzed (Participants) | 25 | 26
h*ng/mL | 2458.4 (28.2) | 2821.8 (34.3)
Statistical Analysis 1: Comparison: Sitravatinib Malate Salt Capsule vs Sitravatinib Free Base Capsule; [analysis description as in outcome 1, analysis 1]; Test type: Other; Ratio of Geometric Least Squares Means = 87.50, 90% CI 2-sided [78.12 to 98.01]

3. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of Sitravatinib
Time Frame: Predose and 0.5, 1, 2, 4, 6, 8, 12, 24, 48, 72 and 168 hours postdose in each study period
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Sitravatinib Malate Salt Capsule | Sitravatinib Free Base Capsule
Number analyzed (Participants) | 25 | 26
ng/mL | 54.96 (32.9) | 62.40 (37.7)
Statistical Analysis 1: Comparison: Sitravatinib Malate Salt Capsule vs Sitravatinib Free Base Capsule; [analysis description as in outcome 1, analysis 1]; Test type: Other; Ratio of Geometric Least Squares Means = 88.80, 90% CI 2-sided [77.41 to 101.87]

4. Primary Outcome: Time of the Maximum Observed Plasma Concentration (Tmax) of Sitravatinib
Time Frame: Predose and 0.5, 1, 2, 4, 6, 8, 12, 24, 48, 72 and 168 hours postdose in each study period
Population: as for outcome 1
Measure: Median (Full Range); unit: Hours
Arm/Group | Sitravatinib Malate Salt Capsule | Sitravatinib Free Base Capsule
Number analyzed (Participants) | 25 | 26
Hours | 8.000 [6.00 to 12.02] | 8.000 [6.00 to 12.00]

5. Primary Outcome: Apparent Terminal Elimination Half-life (T1/2) of Sitravatinib
Time Frame: Predose and 0.5, 1, 2, 4, 6, 8, 12, 24, 48, 72 and 168 hours postdose in each study period
Population: as for outcome 1
Measure: Median (Full Range); unit: Hours
Arm/Group | Sitravatinib Malate Salt Capsule | Sitravatinib Free Base Capsule
Number analyzed (Participants) | 25 | 26
Hours | 30.850 [21.24 to 41.88] | 28.490 [22.27 to 39.35]

6. Primary Outcome: Apparent Total Plasma Clearance (CL/F) of Sitravatinib
Time Frame: Predose and 0.5, 1, 2, 4, 6, 8, 12, 24, 48, 72 and 168 hours postdose in each study period
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters/hour
Arm/Group | Sitravatinib Malate Salt Capsule | Sitravatinib Free Base Capsule
Number analyzed (Participants) | 25 | 26
Liters/hour | 39.61 (28.8) | 41.48 (34.5)

7. Primary Outcome: Apparent Volume of Distribution (Vz/F) of Sitravatinib
Time Frame: Predose and 0.5, 1, 2, 4, 6, 8, 12, 24, 48, 72 and 168 hours postdose in each study period
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters
Arm/Group | Sitravatinib Malate Salt Capsule | Sitravatinib Free Base Capsule
Number analyzed (Participants) | 25 | 26
Liters | 1733.8 (28.7) | 1780.6 (35.3)

8. Secondary Outcome: Number of Participants With Adverse Events
Description: Adverse events (AEs) and serious adverse events are defined as an AE that starts during or after the first dose, or starts prior to the first dose and increases in severity after the first dose, including vital signs, physical examination, electrocardiogram, and laboratory parameters
Time Frame: Up to Week 8
Population: Safety Analysis Set included participants who received at least 1 dose of sitravatinib
Measure: Count of Participants; unit: Participants
Groups:
- Sitravatinib Malate Salt Capsule: Sitravatinib malate salt capsule 100 mg on Day 1 of Periods 1 and 2, with a minimum washout period between dose administrations of 14 days
- Sitravatinib Free Base Capsule: Sitravatinib free base capsule 120 mg on Day 1 of Periods 1 and 2, with a minimum washout period between dose administrations of 14 days
Arm/Group | Sitravatinib Malate Salt Capsule | Sitravatinib Free Base Capsule
Number analyzed (Participants) | 25 | 26
Participants
  At least 1 treatment-emergent adverse event (TEAE) | 10 | 8
  Grade 3 or 4 TEAEs | 0 | 0
  Serious adverse events | 0 | 0
  TEAE leading to permanent discontinuation of study treatment | 0 | 1
  TEAE leading to death | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to Week 8
Description: Safety Analysis Set included participants who received at least 1 dose of sitravatinib
Groups:
- Sitravatinib Malate Salt Capsule: Sitravatinib malate salt capsule 100 mg on Day 1 in Periods 1 and 2, with a minimum washout period between dose administrations of 14 days
- Sitravatinib Free Base Capsule: Sitravatinib free base capsule 120 mg (reference) on Day 1 in Periods 1 and 2, with a minimum washout period between dose administrations of 14 days
Arm/Group | Sitravatinib Malate Salt Capsule | Sitravatinib Free Base Capsule
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/26
Other Adverse Events (participants affected / at risk) | 10/25 | 8/26
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sitravatinib Malate Salt Capsule (N=25) | Sitravatinib Free Base Capsule (N=26)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Palatal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Catheter site bruise (General disorders) | 1 (1) | 0 (0)
Catheter site pain (General disorders) | 1 (1) | 1 (1)
Catheter site related reaction (General disorders) | 0 (0) | 1 (1)
Vessel puncture site bruise (General disorders) | 3 (4) | 0 (0)
Vessel puncture site pain (General disorders) | 2 (2) | 0 (0)
Alanine aminotransferase increased (Investigations) | 2 (2) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Lethargy (Nervous system disorders) | 0 (0) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
BeiGene has 18 months from the end of the study at all sites to publish overall study results. After the 1st multi-site publication or the expiration of publication period, Investigators are free to publish/present the results of the study. Investigators must submit all draft publications/presentations to us for review 60 days prior to the planned publication/presentation date. BeiGene may request deletion of its confidential information and may request a further delay to protect its IP rights.

DOCUMENTS (2):
  • Study Protocol (2020-07-12): https://cdn.clinicaltrials.gov/large-docs/50/NCT04472650/Prot_000.pdf
  • Statistical Analysis Plan (2020-09-09): https://cdn.clinicaltrials.gov/large-docs/50/NCT04472650/SAP_001.pdf